CLINICAL TRIAL: NCT03505567
Title: Pilot Comparative Study of the Kowa OCT Bi-μ and the Optovue iVue 100
Brief Title: Study to Compare Kowa OCT Bi-μ and the Optovue iVue 100
Acronym: OCT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Kowa Research Institute, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: RT1-01US
Record Dates: First submitted 2018-04-16; First posted 2018-04-23 (Actual); Last update posted 2018-09-10 (Actual); Status verified 2018-09

CONDITIONS: Glaucoma; Retinal Disease; Healthy
MeSH Terms: conditions — Glaucoma; Retinal Diseases

STUDY DESIGN:
Intervention Model Description: Eligible participants assigned two interventions under random sequence assignments.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

ARMS (1):
- Random Sequenced Interventions (Other): Participants from three condition groups (normal, glaucoma, retinal disease) assigned two interventions (Kowa OCT Bi-μ and the Optovue iVue 100) under random sequence assignments.
  Interventions: Device: KOWA OCT Bi-µ; Device: Optovue iVue 100

INTERVENTIONS:
Device: KOWA OCT Bi-µ — Non-contact, ultra-high resolution ophthalmic imaging system for fundus imaging and axial cross-sectional and three-dimensional imaging of retinal structures.
Device: Optovue iVue 100 — U.S. Food and Drug Administration (FDA) cleared and commercially available Optovue iVue 100

SUMMARY:
This study is a prospective comparative study to gather pilot agreement and precision data in normal subjects, subjects with glaucoma, and subjects with retinal disease.

ELIGIBILITY:
Inclusion Criteria (Normal Group):

* Subjects with normal eye examinations (without pathology other than cataract) in one or both eyes on the date of the study visit;
* Subjects with intraocular pressure (IOP) ≤ 21 mmHg in the normal eye(s) on the date of the study visit; and
* Subjects with current best-spectacle-corrected visual acuity (BSCVA) of 20/40 or better in the normal eye(s) on the date the study visit.

Exclusion Criteria (Normal Group):

* Subjects unable to tolerate ophthalmic imaging;
* Subjects with ocular media not sufficiently clear to obtain acceptable OCT images;
* Subjects with any current ocular pathology other than cataract in the normal eye(s), as determined by self-report and/or investigator assessment at the study visit;
* Subjects with current narrow anterior chamber drainage angle in the normal eye(s), as determined by self-report and/or investigator assessment at the study visit; and
* Subjects with a history of leukemia, dementia or multiple sclerosis.

Inclusion Criteria (Glaucoma Group):

* Subjects who have been diagnosed with glaucoma in the glaucoma study eye(s), with optic nerve damage as evidenced by either of the following optic disc or retinal nerve fiber layer structural abnormalities observed via fundus exam during the study visit:

  1. Diffuse thinning, focal narrowing, or notching of the optic disc rim, especially at the inferior or superior poles with or without disc hemorrhage; or
  2. Optic disc neural rim asymmetry of the two eyes consistent with loss of neural tissue;
* Subjects with a current BSCVA of 20/40 or better in the glaucoma study eye(s) on the date of the visit; and
* History of visual field defects within the previous two (2) months from the study visit or measured on the day of the study visit that is consistent with glaucomatous optic nerve damage based on at least one of the following findings:

  1. On pattern deviation (PD), there exists a cluster of 3 or more points in an expected location of the visual field depressed below the 5% level, at least 1 of which is depressed below the 1% level; and
  2. Glaucoma hemi-field test "outside normal limits."

Exclusion Criteria (Glaucoma Group):

* Subjects unable to tolerate ophthalmic imaging;
* Subjects with ocular media not sufficiently clear to obtain acceptable OCT images;
* Subjects with at least one Humphrey Field Analyzer (HFA) visual field (24-2 SITA Standard, white on white) measured on the day of the study visit, or within the previous two (2) months from the study visit with unreliable results, defined as fixation losses > 20%, or false positives > 33%, or false negatives > 33% in the glaucoma study eye(s);
* Subjects with any current ocular pathology except glaucoma in the glaucoma study eye(s), as determined by self-report and/or investigator assessment on the day of the study visit; and
* Subjects with a history of leukemia, dementia or multiple sclerosis.

Inclusion Criteria (Retinal Disease Group):

* Subjects with current IOP ≤ 21 mmHg in the retinal disease study eye(s) on the day of the study visit;
* Subjects with a current BSCVA of 20/400 or better in the retinal disease study eye(s) at the study visit; and
* Subjects diagnosed with retinal pathology including but not limited to: Macular Degeneration, Diabetic Macular Edema, Diabetic Retinopathy, Macular Hole, Epiretinal Membrane, Cystoid Macular Edema, and others in the retinal disease study eye(s) as confirmed within the past six (6) months.

Exclusion Criteria (Retinal Disease Group):

* Subjects unable to tolerate ophthalmic imaging;
* Subjects with ocular media not sufficiently clear to obtain acceptable OCT images;
* Subjects with glaucoma or any ocular pathology other than retinal pathology (e.g. cornea pathology) in the retinal disease study eye(s), as determined by self-report and/or investigator assessment at the study visit;
* Subjects with current narrow anterior chamber drainage angle in the retinal disease study eye(s), as determined by self-report and/or investigator assessment at the study visit; and
* Subjects with a history of leukemia, dementia or multiple sclerosis.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2018-04-21 (Actual); Primary Completion 2018-09-01 (Actual); Study Completion 2018-09-01 (Actual)

PRIMARY OUTCOMES:
Compare KOWA OCT Bi-μ and Optovue iVue 100 | 1-2 days
  1. Full retinal thickness [Early Treatment Diabetic Retinopathy Study (ETDRS) Grid]
  2. Full retinal thickness (Manual Measurement)
  3. Retinal nerve fiber layer thickness
  4. Ganglion cell complex thickness
  5. Full retinal thickness map

SECONDARY OUTCOMES:
Safety: Evaluate any adverse events found during the clinical study | 1-2 days
  Evaluate any adverse events found during the clinical study

CONTACTS AND LOCATIONS:
Overall Officials: David Hosford, MD, Ph.D, Study Director — Kowa Research Institute, Inc.
Locations (1):
- Andover Eye Associates, Andover, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No